CLINICAL TRIAL: NCT00005983
Title: Randomized Trial of Post-Mastectomy Radiotherapy in Stage II Breast Cancer in Women With One to Three Positive Axillary Nodes Phase III
Brief Title: S9927 Radiation Therapy After Surgery, Chemotherapy, and/or Hormone Therapy in Stage II Breast Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: due to lack of accrual
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH); North Central Cancer Treatment Group (Network); American College of Surgeons (Other); Eastern Cooperative Oncology Group (Network); Radiation Therapy Oncology Group (Network); Cancer and Leukemia Group B (Network); NCIC Clinical Trials Group (Network); NSABP Foundation Inc (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000067971; U10CA032102 (NIH); S9927 (Other: SWOG); S9927 (Other: ACOSOG); CAN-NCIC-MA25 (Other: NCIC-CTG); CLB-49910 (Other: CALGB); S9927 (Other: ECOG); S9927 (Other: NCCTG); S9927 (Other: NSABP); RTOG-9915 (Other: RTOG)
Record Dates: First submitted 2000-07-05; First posted 2003-01-27 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- surgery (Active Comparator): surgery followed by observation
  Interventions: Procedure: surgery
- surgery followed by RT (Experimental): Surgery followed by radiation therapy
  Interventions: Radiation: radiation therapy; Procedure: surgery

INTERVENTIONS:
Radiation: radiation therapy
  Arms: surgery followed by RT
Procedure: surgery — surgery

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. It is not yet known whether mastectomy, chemotherapy, and/or hormone therapy are more effective with or without radiation therapy in treating breast cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of mastectomy, chemotherapy, and/or hormone therapy with or without radiation therapy in treating women who have stage II breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare overall and disease-free survival in women with stage II breast cancer with one to three positive nodes treated with radiotherapy vs observation only after mastectomy and adjuvant chemotherapy and/or hormonal therapy.
* Compare local regional control in patients treated with these regimens.
* Assess the potential toxic effects of radiotherapy in this patient population.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to prior systemic hormonal therapy (chemotherapy with or without hormonal therapy vs hormonal therapy alone), prior taxane exposure (yes vs no), and duration of chemotherapy (no chemotherapy vs less than 3 months vs 3-5 months vs 6 months or more). Patients are randomized to one of two treatment arms.

* Arm I: Patients undergo radiotherapy 5 days a week for 5 weeks.
* Arm II: Patients are observed for disease progression. Patients are followed every 6 months for 2 years and then annually for 15 years.

PROJECTED ACCRUAL: A total of 2,500 patients (1,250 per treatment arm) will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage II adenocarcinoma of the breast (T1-2, N1, M0)

  * Primary tumor no greater than 5 cm
  * At least 1 but no more than 3 positive axillary lymph nodes
  * Nodes cannot be positive solely by cytokeratin staining
  * No apocrine, adenocystic, or squamous cell carcinomas or sarcomas of the breast
  * No bilateral breast cancer
  * No active local regional disease
* Must have undergone a modified radical mastectomy with a level I and II with or without a level III axillary dissection (at least 10 nodes examined) within the past 8 months

  * Surgical margins negative for invasive and noninvasive ductal carcinoma
  * No gross extracapsular disease or residual disease in the axilla
  * Microscopic extracapsular extension allowed
* No mastectomy after local failure following lumpectomy
* Must have received adjuvant chemotherapy and/or hormonal therapy after mastectomy
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 21 and over

Sex:

* Female

Menopausal status:

* Pre- or post-menopausal

Performance status:

* Zubrod 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No other prior malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No serious medical or psychiatric illness that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior trastuzumab (Herceptin)

Chemotherapy:

* See Disease Characteristics
* No more than 6 weeks since prior adjuvant chemotherapy
* No other prior chemotherapy
* Concurrent adjuvant chemotherapy allowed

Endocrine therapy:

* See Disease Characteristics
* Concurrent adjuvant hormonal therapy allowed

Radiotherapy:

* No prior chest wall or nodal radiotherapy

Surgery:

* See Disease Characteristics
* Breast reconstruction allowed

Other:

* Concurrent registration on another adjuvant chemotherapy or hormonal therapy study is allowed

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2000-06; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lori J. Pierce, MD, Study Chair — University of Michigan Rogel Cancer Center; Michael G. Haddock, MD, Study Chair — Mayo Clinic; Stephen B. Edge, MD, Study Chair — Roswell Park Cancer Institute; Eric A. Strom, MD, FACR, Study Chair — M.D. Anderson Cancer Center; Lawrence J. Solin, MD, FACR, Study Chair — Abramson Cancer Center at Penn Medicine; Lawrence B. Marks, MD, Study Chair — Duke University; Timothy J. Whelan, MD, Study Chair — Margaret and Charles Juravinski Cancer Centre; Melvin Deutsch, MD, Study Chair — UPMC Cancer Center at UPMC Presbyterian
Locations (1):
- Cancer Care Ontario-Hamilton Regional Cancer Centre, Hamilton, Ontario, Canada